CLINICAL TRIAL: NCT03500809
Title: Efficacy and Safety of Aqueous Humour Release (Burping) Performed at the Slit-lamp to Treat Acute Intraocular Pressure (IOP) Spikes Post-cataract Surgery
Brief Title: Aqueous Release to Treat IOP Spikes Post-cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bedford Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Anant Sharma, Consultant Ophthalmic Surgeon, Bedford Hospital NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 240539
Record Dates: First submitted 2018-04-06; First posted 2018-04-18 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Post-Op Complication; Raised Ocular Pressure
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aqueous release (Burping) of the wound (Experimental): Following uneventful cataract surgery, wound "burping" will be performed in all eligible patients who gave their informed consent. The procedure will be offered whenever the intraocular pressure (IOP) is either higher than 30 mmHg or deemed inappropriate in view of the ocular condition (e.g. glaucoma).
  After 'burping' the wound, patients will have their IOP measured using Goldmann application tonometry (GAT) immediately and at 2 hours. The 'burping' procedure will be repeated until satisfactory pressure is achieved and care will be taken to avoid shallowing of the anterior chamber while fluid is released. We will assess for the presence of leaks from the wound with a Seidel test with fluorescein 5% once the IOP is satisfactory. To prevent any infection after each procedure, we will prescribe post-op drops including chloramphenicol 0.5% four times a day for 2 weeks or minimum of 3 days and these will continue as per routine. All other complications will be recorded at follow-up.
  Interventions: Procedure: Aqueous release of the wound

INTERVENTIONS:
Procedure: Aqueous release of the wound — 1. Anaesthetic drop (tetracaine 1%) followed by povidone iodine 5% drop is instilled. After 5 minutes, a sterile 30 gauge needle tip is pressed on the posterior lip of the one of the existing cuts (paracentesis or main wound) from cataract surgery to release the fluid and consequently the pressure.
  2. This will be performed under careful monitoring to avoid any undesirable shallowing of the anterior chamber of the eye.
  Other Names: 'Burping' procedure

SUMMARY:
Intraocular pressure (IOP) rise after cataract surgery is an important and common problem. Over 300,000 cataract operations are done per year in the United Kingdom alone. IOP rise can adversely affect vision and can be particularly detrimental in glaucoma patients with pre-existing visual field defects. The aim of this study is to evaluate the efficacy and safety of aqueous humor release (also known as burping of the wound), a procedure that has been used for decades to quickly reduce acute IOP spikes following cataract surgery.

Currently there is no published evidence on a standard technique to perform wound burping. Similarly there is uncertainty around the amount and duration of the IOP decrease, and the type and frequency of complications eventually associated. This will be the first research project formally evaluating this procedure. This study will also help allay issues over fluid release in high IOPs and consequences of such dramatic IOP drop which concerns ophthalmologists who do not routinely use this technique.

DETAILED DESCRIPTION:
At present there is no de facto standard to manage acute intraocular pressure (IOP) rise following cataract surgery. Several drugs, both topical and systemic, have been tested for their ability to blunt the acute IOP spike, nevertheless none has proven to be superior and consistently effective. Oral acetazolamide has demonstrated to help controlling IOP spikes following cataract surgery in glaucomatous eyes. However there are still constraints in its widespread use, as it may be contraindicated in patients with poor renal function, sickle cell disease and sulpha drug allergy.

As a result, many units including Moorfields Eye Hospital have used a technique called known as 'burping of the corneal wound' to release fluid from inside the anterior chamber of the eye. This makes logical sense as it reduces the pressure immediately and may remove some of the causes for raised IOP such as retained viscoelastic and inflammatory molecules from inside the eye. This technique has also been used to reduce IOP in patients already receiving pharmaceutical treatment.

The technique has been used for decades, however, there is no published evidence of a proposed technique, range of IOP decrease or frequency of complications. Thus, most surgeons in most units are cautious of 'burping the wound' as it may induce infection or other complications compromising the surgical outcome due to the sudden reduced IOP reduction. Nevertheless a similar approach, needle penetrating the eye to release aqueous and reduce IOP, is becoming more popular as the first approach to treat an acute angle closure crisis, where the presenting IOP is often very high, i.e. a much more difficult and dangerous situation than post cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose post-operative IOP was regarded to be too high for visual safety, or higher than 30mmHg, on the same day or within 1 week of the surgery

Exclusion Criteria:

* Patients with IOP less than 30 mmHg or IOP deemed by clinician not too high to treat
* Patients unable to cooperate
* Patients who have undergone complicated cataract surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-12 (Estimated); Primary Completion 2019-01-12 (Estimated); Study Completion 2019-07-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 'burping' the wound to reduce IOP (mmHg) post-cataract surgery when measured using Goldmann application tonometry (GAT) | 6 months
  Reduction in IOP (mmHg) post-cataract surgery after the 'burping' procedure

SECONDARY OUTCOMES:
Range of IOP decrease (mmHg) | 6 months
  To observe and record the range of IOP decrease (mmHg) from individual 'burping' procedures
Frequency of complications post-'burping' procedure | 6 months
  Observing the frequency of complications, including but not limited to, severe pain, worsening of vision, or infection

CONTACTS AND LOCATIONS:
Overall Officials: Anant Sharma, MBBS, FRCOphth, Principal Investigator — Bedford Hospital Moorfields Eye Unit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Day AC, Donachie PH, Sparrow JM, Johnston RL; Royal College of Ophthalmologists' National Ophthalmology Database. The Royal College of Ophthalmologists' National Ophthalmology Database study of cataract surgery: report 1, visual outcomes and complications. Eye (Lond). 2015 Apr;29(4):552-60. doi: 10.1038/eye.2015.3. Epub 2015 Feb 13. PMID 25679413
- [Background] Kim JY, Jo MW, Brauner SC, Ferrufino-Ponce Z, Ali R, Cremers SL, Henderson BA. Increased intraocular pressure on the first postoperative day following resident-performed cataract surgery. Eye (Lond). 2011 Jul;25(7):929-36. doi: 10.1038/eye.2011.93. Epub 2011 Apr 29. PMID 21527959
- [Background] Tranos P, Bhar G, Little B. Postoperative intraocular pressure spikes: the need to treat. Eye (Lond). 2004 Jul;18(7):673-9. doi: 10.1038/sj.eye.6701319. PMID 15002028
- [Background] Kass MA, Gordon MO, Gao F, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JK, Miller JP, Parrish RK, Wilson MR; Ocular Hypertension Treatment Study Group. Delaying treatment of ocular hypertension: the ocular hypertension treatment study. Arch Ophthalmol. 2010 Mar;128(3):276-87. doi: 10.1001/archophthalmol.2010.20. PMID 20212196
- [Background] Hayashi K, Yoshida M, Manabe SI, Yoshimura K. Prophylactic Effect of Oral Acetazolamide against Intraocular Pressure Elevation after Cataract Surgery in Eyes with Glaucoma. Ophthalmology. 2017 May;124(5):701-708. doi: 10.1016/j.ophtha.2016.12.027. Epub 2017 Jan 19. PMID 28110949
- [Background] Wang Q, Harasymowycz P. Short-Term Intraocular Pressure Elevations after Combined Phacoemulsification and Implantation of Two Trabecular Micro-Bypass Stents: Prednisolone versus Loteprednol. J Ophthalmol. 2015;2015:341450. doi: 10.1155/2015/341450. Epub 2015 Jul 21. PMID 26266045
- [Background] Cioboata M, Anghelie A, Chiotan C, Liora R, Serban R, Cornacel C. Benefits of anterior chamber paracentesis in the management of glaucomatous emergencies. J Med Life. 2014;7 Spec No. 2(Spec Iss 2):5-6. PMID 25870663